CLINICAL TRIAL: NCT01485666
Title: Reduce Driveline Trauma Through Stabilization and Exit Site Management (RESIST) Pilot Study Protocol
Brief Title: Thoratec's Reduce Driveline Trauma Through Stabilization and Exit Site Management Study
Acronym: RESIST
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TC06072011-1
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Left Ventricular Assist Device; Percutaneous Lead Management
Keywords: Thoratec; HeartMate II; heart-assist devices; driveline or percutaneous lead management; HeartMate II Percutaneous Lead Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Percutaneous Lead Management Kit — A kit of commercially available components to be used for HeartMate II driveline exit site cleaning, dressing and stabilization
  Other Names: Thoratec; HeartMate II

SUMMARY:
The purpose of this study is to evaluate the feasibility of a Percutaneous Lead Management Kit for HeartMate II driveline stabilization and exit site management.

DETAILED DESCRIPTION:
The Percutaneous Lead Management Kit is a combination of commercially available components that are packaged together in a kit to be used for HeartMate II driveline exit site cleaning, dressing and stabilization. The RESIST study is a prospective, non-randomized study to evaluate the wearability and usability of the Percutaneous Lead Management Kit. Evaluation of the Percutaneous Lead Management Kit for wearability and usability will be performed for 30 days from enrollment. Study patients will also be followed for up to 6 months for any evidence of driveline infection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* 16 years of age or older
* Supported by HeartMate II LVAD continuously for at least 6 months and not currently hospitalized
* Will continue on LVAD support for at least another 30 days
* No driveline or systemic infection
* Willing and able to perform kit dressing changes at least once every 7 days for 30 days
* Can fill out study forms
* Can use a digital camera
* Willing to return to clinic for final study visit in 30 days

Exclusion Criteria:

* High risk for non-compliance
* Ongoing mechanical circulatory support other than HeartMate II LVAD
* Sensitivity to kit components
* Skin condition that may react to kit component adhesives
* Already using all components of Percutaneous Lead Management Kit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ventricular Assist Device clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Demonstration of the wearability and usability of the Percutaneous Lead Management Kit | Up to 30 days

SECONDARY OUTCOMES:
Incidence of adverse reactions to any Percutaneous Lead Management Kit components | Up to 6 months
Evidence of driveline infection | Up to 6 months
Durability of the Percutaneous Lead Management Kit's infection mitigation and stabilization | Up to 7 days continuous kit use

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec Corporation
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sharp Memorial Hospital, San Diego, California
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina